CLINICAL TRIAL: NCT02091440
Title: Clinical Evaluation of the HW005 Ventricular Assist System for the Treatment of Advanced Heart Failure
Brief Title: Clinical Evaluation of HW005 Ventricular Assist System for the Treatment of Advanced Heart Failure in Japan
Acronym: HW005
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HW005/ Japan
Record Dates: First submitted 2014-03-17; First posted 2014-03-19 (Estimated); Results first posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-07

CONDITIONS: Heart Failure
Keywords: Medical Device; Thoracic Surgical Procedure; Pumps Heart Assist; Ventricular Assist Device
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HW005 Ventricular Assist System (Other): Implant of the HW005 Ventricular Assist System.
  Interventions: Device: Implant of the HW005 Ventricular Assist System.

INTERVENTIONS:
Device: Implant of the HW005 Ventricular Assist System. — The HW005 Pump is in implantable centrifugal pump that was designed to provide flows up to 10 L/min. It is a small device which is both lightweight and simple to use.

SUMMARY:
The purpose of the study is to evaluate the safety and effectiveness of the HW005 System in patients listed for cardiac transplantation with refractory, advanced heart failure at risk of death.

DETAILED DESCRIPTION:
The primary endpoint is success at 180 days which is expressed as a simple proportion and defined as alive on the originally implanted HW005 or transplanted or explanted for recovery. Patients must survive 60 days post-explant for recovery to be considered successful. The primary endpoint is not statistically powered. The six eligible implanted cases will be evaluated as a proportion of success accompanied by a 95% exact confidence interval and presented alongside the ADVANCE results for visual comparison.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with irreversible end-stage heart failure of New York Heart Association (NYHA) class III or IV and a history of class IV who are eligible for heart transplantation.
2. Patients who are dependent on medication of inotropes or intra-aortic balloon pump (IABP).
3. Body Surface Area (BSA) ≥1.2 m2. In addition other factors may be taken into consideration, including chest size, abdominal fat (lack of abdominal fat may preclude a pump pocket) and any other physical characteristics that might be benefited by an intra-pericardial pump in a small person.
4. Patients who are aged less than 65 years of age.
5. Patients must be able to understand the limits and complications associated with the HW005 Ventricular Assist System.
6. Female patients of childbearing potential must agree on contraception for the duration of the study.
7. The patient or the legal representative has signed the informed consent form.

Exclusion Criteria:

1. Severe illness other than heart disease which would exclude cardiac transplantation.
2. Inadequate family/social support.
3. Active, uncontrolled infection despite appropriate antibiotic, antiviral or antifungal treatment.
4. Existence of any ongoing mechanical circulatory support (MCS) other than an IABP.
5. Prior cardiac transplant or cardiomyoplasty.
6. Acute myocardial infarction within 14 days of implant.
7. Uncorrected thrombocytopenia or generalized coagulopathy.
8. Intolerance to anticoagulant or antiplatelet therapies or any other peri- or postoperative therapy that the investigator may administer based upon the patient's health status.
9. Patients for whom the use of a left ventricular assist device (LVAD) is contraindicated due to an ongoing aortic/cardiac aneurysm, intraventricular septum rupture and/or use of a mechanical heart valve.
10. Etiology of heart failure is due to, or associated with, uncorrected thyroid disease, obstructive cardiomyopathy, pericardial disease, amyloidosis, active myocarditis or restrictive cardiomyopathy.
11. Patients with irreversible hepatic dysfunction.
12. Patients with irreversible renal dysfunction.
13. Pregnancy.
14. Patients with serious chronic obstructive pulmonary disease (COPD) (Forced Expiratory Volume in the first second (FEV1) < 50%).
15. Pulmonary vascular resistance is unresponsive (fixed) to pharmacologic manipulation as demonstrated by a pulmonary artery systolic pressure exceeding 60mmHg in conjunction with any one of the two following variables:

    * Pulmonary vascular resistance is greater than 6 Woods Units or
    * Transpulmonary gradient exceeds 15 mmHg
16. Cardiothoracic surgery within 14 days of implantation.
17. Peripheral vascular disease with rest pain or ischemic ulcers of the extremities.
18. Pulmonary embolus within three weeks of enrollment as documented by computed tomography (CT) scan or nuclear scan.
19. Patients have moderate to severe aortic insufficiency without plans for correction during pump implantation surgery. Correction may include aortic valve repair at the time of implant.
20. The patient who has advanced calcification in the ascending aorta and/or the descending aorta.
21. Serious right heart failure as defined by the anticipated need for right ventricular assist device (RVAD) support or extracorporeal membrane oxygenation (ECMO) at the time of screening.
22. Patients with severe central nervous system disorder or severe cerebral vascular disorder.
23. Patients with a history of drug intoxication, alcohol dependence.
24. Patients unwilling or unable to comply with study requirements.
25. Patients who refuse transfusion.
26. Patients who in the investigator judgement are deemed to be unsuitable as a subject.
27. Patients who are participating in another clinical trial involving investigational drugs or devices.

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-03; Primary Completion 2015-03 (Actual); Study Completion 2018-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoshiki Sawa, MD, Principal Investigator — Osaka University Hospital
Locations (5):
- Japan (5):
  - Kyushu University Hospital, Fukuoka, Kyushu
  - Tohoku University Hospital, Sendai, Tohoku
  - Osaka University Hospital, Osaka
  - National Cerebral and Cardiovascular Center Hospital, Osaka
  - The University of Tokyo Hospital, Tokyo

RESULTS

PARTICIPANT FLOW:
Groups:
- HW005 Ventricular Assist System: Implant of the HW005 Ventricular Assist System.: The HW005 Pump is an implantable centrifugal pump that was designed to provide flows up to 10 L/min. It is a small device which is both lightweight and simple to use.
Period: Overall Study
Arm/Group | HW005 Ventricular Assist System
Started | 6
Primary Endpoint (Success at 180 Days) | 6
Overall Survival at 180 Days | 6
Completed | 4
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | HW005 Ventricular Assist System
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Japan | 6
New York Heart Association (NYHA) Classification [Count of Participants; unit: Participants] — The New York Heart Association (NYHA) Functional Classification places patients with heart failure in one of four categories based on how much they are limited during physical activity.
  Class I (best): No limitation of physical activity.
  Class II: Slight limitation of physical activity. Comfortable at rest.
  Class III: Marked limitation of physical activity. Comfortable at rest.
  Class IV (worst): Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest.
  Participants
    Class I | 0
    Class II | 0
    Class III | 3
    Class IV | 3
Six-Minute Walk Test [Mean (Standard Deviation); unit: meters] | 135.8 (160.12)
Kansas City Cardiomyopathy Questionnaire (KCCQ) scores [Mean (Standard Deviation); unit: units on a scale] — The KCCQ is a self-evaluation questionnaire for patients with heart failure to assess the severity of their symptoms how it may affect their lives. All scores range between 0 (worst) - 100 (best).
  For example: Social Limitation score of 100 means no social limitation at all
  Total Symptom Score: mean of Symptom Frequency and Symptom Burden scores
  Overall Summary Score: mean of Physical Limitation, Symptom Stability, Total Symptom, Quality of Life and Social Limitation scores
  Clinical Summary Score: mean of Physical Limitation and Total Symptom scores
  units on a scale
    KCCQ Physical Limitation | 45.0 (31.69)
    KCCQ Symptom Stability | 37.5 (26.22)
    KCCQ Self-Efficacy | 75.0 (22.36)
    KCCQ Quality of Life | 31.9 (27.09)
    KCCQ Social Limitation | 9.4 (13.26)
    KCCQ Overall Summary Score | 45.5 (28.44)
    KCCQ Clinical Summary Score | 56.4 (33.89)
    KCCQ Symptom Frequency | 66.0 (39.91)
    KCCQ Symptom Burden | 69.4 (38.97)
    KCCQ Total Symptom Score | 67.7 (39.32)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Alive on the Implanted HW005 Ventricular Assist System or Transplanted or Explanted for Recovery at 180 Days
Description: The primary endpoint is success at 180 days which is defined as alive on the originally implanted HW005 Ventricular Assist System or transplanted or explanted for recovery. Patients must survive 60 days post-explant for recovery to be considered successful.
Time Frame: 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | HW005 Ventricular Assist System
Number analyzed (Participants) | 6
Participants | 6
Statistical Analysis 1: Comparison: HW005 Ventricular Assist System; Test type: Other — Single group; Proportion = 100

2. Secondary Outcome: Number of Participants Alive on the Implanted HW005 Ventricular Assist System at 180 Days
Time Frame: 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | HW005 Ventricular Assist System
Number analyzed (Participants) | 6
Participants | 6
Statistical Analysis 1: Comparison: HW005 Ventricular Assist System; Test type: Other — Single group; Kaplan-Meier Survival = 100

3. Secondary Outcome: Incidence of All Serious Adverse Events (SAEs) and Unanticipated Adverse Device Effects (UADEs)
Description: SAEs are defined as events that result in death, are life-threatening, result in permanent disability, require medical treatment to prevent permanent disability or require surgical intervention or hospitalization.
  UADEs are defined as any serious adverse device effect which by its nature, incidence, severity or outcome has not been identified in the current version of the risk analysis report.
  Events were categorized using the Japanese registry for Mechanically Assisted Circulatory Support (J-MACS) definitions.
Time Frame: Through study completion, an average of 44.5 months
Measure: Number; unit: event rate per patient year
Arm/Group | HW005 Ventricular Assist System
Number analyzed (Participants) | 6
event rate per patient year
  J-MACS SAEs | 1.24
  UADEs | 0
Statistical Analysis 1: Comparison: HW005 Ventricular Assist System; Test type: Other — Single group; Incidence = 1.24

4. Secondary Outcome: Incidence of All Device Failures and Device Malfunctions.
Description: The device failures and malfunctions are the failures on pumping function due to thrombosis inside/outside of the implanted pump, the mechanical failures of the implanted components, the mechanical failures of the external components and the failures due to the user.
  Events were categorized using the J-MACS definitions.
Time Frame: Through study completion, an average of 44.5 months
Measure: Number; unit: event rate per patient year
Arm/Group | HW005 Ventricular Assist System
Number analyzed (Participants) | 6
event rate per patient year | 1.66
Statistical Analysis 1: Comparison: HW005 Ventricular Assist System; Test type: Other — Single group; Incidence = 1.66

5. Secondary Outcome: Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) Quality of Life Score at 6 and 24 Months
Description: The KCCQ is a self-evaluation questionnaire for patients with heart failure to assess the severity of their symptoms how it may affect their lives. Scores range between 0 (worst) - 100 (best).
  Values in the table were calculated as the value at Month 6 (180 days) minus Screening and at Month 24 (after FU completion) minus Screening.
  The positive change in KCCQ score indicates an improvement in patient Quality of Life.
Time Frame: Screening, Month 6 (180 days) and Month 24 (after follow-up (FU) completion)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HW005 Ventricular Assist System
Number analyzed (Participants) | 6
score on a scale
  Month 6 | 22.2 (12.55)
  Month 24 | 19.4 (11.39)
Statistical Analysis 1: Comparison: HW005 Ventricular Assist System; Test type: Other — Single group; Change from baseline = 19.4, 95% CI 2-sided [7.5 to 31.4], Standard Deviation 11.39 — Confidence interval based on t-distribution

6. Secondary Outcome: Change in NYHA Patient Classification (Patient Functional Status) at 6 and 24 Months
Description: The New York Heart Association (NYHA) Functional Classification places patients with heart failure in one of four categories based on how much they are limited during physical activity.
  Class I (best): No limitation of physical activity.
  Class II: Slight limitation of physical activity. Comfortable at rest.
  Class III: Marked limitation of physical activity. Comfortable at rest.
  Class IV (worst): Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest.
  A shift from a higher class (e.g. Class IV) to a lower class (e.g. Class II) indicates an improvement in patient health and functional status.
Time Frame: Screening, Month 6 (180 days) and Month 24 (after FU completion)
Measure: Count of Participants; unit: Participants
Arm/Group | HW005 Ventricular Assist System
Number analyzed (Participants) | 6
Participants
  Screening: Class I | 0
  Screening: Class II | 0
  Screening: Class III | 3
  Screening: Class IV | 3
  Month 6: Class I | 1
  Month 6: Class II | 5
  Month 6: Class III | 0
  Month 6: Class IV | 0
  Month 24: Class I | 2
  Month 24: Class II | 3
  Month 24: Class III | 1
  Month 24: Class IV | 0
Statistical Analysis 1: Comparison: HW005 Ventricular Assist System; Test type: Other — Single group; Percentage change = -83.33 — Percentage change from 24 months to screening in NYHA classes III and IV. Percentage change is 16.67% - 100% = -83.33%

7. Secondary Outcome: Change in Patient 6-minute Walk Distance (Patient Functional Status) at 6 and 24 Months
Description: For the 6-minute walk test, the patient is asked to walk for 6 minutes. The total distance walked is measured.
  Values in the table were calculated as the value at Month 6 (180 days) minus Screening and at Month 24 (after FU completion) minus Screening.
  A positive change in 6-minute walk distance indicates an improvement in health and functional status.
Time Frame: Screening, Month 6 (180 days) and Month 24 (after FU completion)
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | HW005 Ventricular Assist System
Number analyzed (Participants) | 6
Meters
  Month 6 | 198.2 (217.01)
  Month 24 | 130.0 (275.32)
Statistical Analysis 1: Comparison: HW005 Ventricular Assist System; Test type: Other — Single group; Change from baseline = 130.0, 95% CI 2-sided [-158.9 to 418.9], Standard Deviation 275.32 — Confidence interval based on t-distribution

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 44.5 months
Arm/Group | HW005 Ventricular Assist System
All-Cause Mortality (participants affected / at risk) | 2/6
Serious Adverse Events (participants affected / at risk) | 5/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HW005 Ventricular Assist System (N=6)
Bleeding requiring re-hospitalization (Injury, poisoning and procedural complications) | 2 (2)
Bleeding requiring re-operation (Injury, poisoning and procedural complications) | 2 (2)
Ventricular Cardiac Arrhythmia (Cardiac disorders) | 2 (2)
Supraventricular Cardiac Arrhythmia (Cardiac disorders) | 2 (3)
Sepsis (Infections and infestations) | 1 (2)
Driveline Exit Site Infection (Infections and infestations) | 1 (1)
Hemorrhagic Cerebrovascular Accident (Vascular disorders) | 1 (3)
Pericardial Fluid Collection (Cardiac disorders) | 2 (2)
Chronic Renal Dysfunction (Renal and urinary disorders) | 1 (1)
Respiratory Dysfunction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Right Heart Failure requiring inotropic therapy (Cardiac disorders) | 1 (2)
Other (General disorders) | 3 (5)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HW005 Ventricular Assist System (N=6)
Bleeding requiring re-hospitalization (Injury, poisoning and procedural complications) | 2 (2)
Bleeding requiring re-operation (Injury, poisoning and procedural complications) | 2 (2)
Ventricular Cardiac Arrhythmia (Cardiac disorders) | 3 (3)
Supraventricular Cardiac Arrhythmia (Cardiac disorders) | 3 (4)
Device Malfunction/Failure (Product Issues) | 2 (5)
Sepsis (Infections and infestations) | 1 (2)
Driveline Exit Site Infection (Infections and infestations) | 2 (2)
Hemorrhagic Cerebrovascular Accident (Vascular disorders) | 1 (3)
Pericardial Fluid Collection (Cardiac disorders) | 2 (2)
Acute Renal Dysfunction (Renal and urinary disorders) | 1 (1)
Chronic Renal Dysfunction (Renal and urinary disorders) | 1 (1)
Respiratory Dysfunction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Right Heart Failure requiring inotropic therapy (Cardiac disorders) | 1 (2)
Other (General disorders) | 6 (86)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI cannot disclose the trial results without the sponsor's permission. The disclosure restriction is not limited by a set period.